CLINICAL TRIAL: NCT00376740
Title: Phase 3 Study of the Effect of Zoledronic Acid in the Prevention of Osteoporosis in Early Breast Cancer Patients Receiving the Aromatase Inhibitor, Letrozole, in the Adjuvant Setting
Brief Title: Effectiveness of Zoledronic Acid in the Prevention of Osteoporosis in Early Breast Cancer Patients Receiving Letrozole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, David B. Geffen, Director of the Oncology Ambulatory Care Clinic, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sor440006ctil
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: breast cancer, postmenopausal, letrozole, zoledronic acid, adjuvant,bone mineral density
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate zoledronic acid (Experimental): Patients on this arm will receive zoledronic acid every 6 months during 2.5 years of letrozole therapy starting within 3 months of the start of letrozole therapy. (5 doses of zoledronic acid)
  Interventions: Drug: zoledronic acid
- Delayed zoledronic acid (Active Comparator): Patients on this arm will receive zoledronic acid during the 2.5 years of letrozole treatment only after the T-score on bone mineral density testing falls below minus 2.0.
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — Zoledronic acid 4 mg IV every 6 months up to 2.5 years after the start of letrozole treatment.
  Other Names: Zomera, zolendronate

SUMMARY:
The purpose of this study is to determine whether zoledronic acid given intravenously every 6 months can prevent reduction in bone mineral density in women with early stage breast cancer receiving adjuvant therapy with the aromatase inhibitor drug letrozole, after having received adjuvant tamoxifen.

DETAILED DESCRIPTION:
Letrozole is an aromatase inhibitor used in the treatment of hormone receptor positive metastatic breast cancer in postmenopausal women.It has more recently been approved for use in many countries as adjuvant therapy for early breast cancer; and is often used in an adjuvant regimen following 2-3 years of tamoxifen treatment or as an extended adjuvant therapy after up to 5 years of tamoxifen. Letrozole inhibits the conversion of androgens to estrogens in vitro and in vivo. Plasma levels of estradiol and related estrogen compounds in postmenopausal patients receiving letrozole are suppressed up to 95% from baseline and are often undetectable.The estrogen deprivation in women receiving letrozole may cause increased bone resorption and bone loss.Studies comparing tamoxifen and aromatase inhibitors, in adjuvant therapy have shown an increase fracture rate, and decreased bone mineral density in patients receiving aromatase inhibitors. Zoledronic acid is an intravenously administered bisphosphonate that inhibits osteoclastic bone resorption. Intravenous bisphosphonates are effective in reducing the rate of skeletal complications, including fractures, in patients with metastatic breast cancer and other tumors when given every few weeks. Small clinical trials have given some evidence that osteoporosis can be effectively treated by one or two doses of intravenous zoledronic acid per year. This study will determine the effect of giving zoledronic acid every 6 months on the bone mineral density of patients receiving letrozole as adjuvant therapy for early breast cancer after having received adjuvant tamoxifen for at least 2.5 years. Patients will be randomized to receive zoledronic acid either at the start of letrozole therapy or when bone mineral density T score drops below - 2 standard deviation or at the occurrence of a non-trauma related fracture.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with histologically documented early (non-metastatic) breast cancer
* Previous treatment with tamoxifen for at least 2.5 years and not more than 3.5 years
* Assigned to receive letrozole treatment
* Karnofsky performance status ≥ 70
* Life expectancy ≥ 16 weeks
* Signed informed consent after full explanation of study by participating clinician and prio to any study specific procedures
* Adjuvant or neoadjuvant chemotherapy is allowed
* No clinical and/or radiologic evidence of distant metastases
* No prior treatment with an aromatase inhibitor
* Able to comply with treatment and scheduled follow-up visits
* Age between 18 and 82 years

Exclusion Criteria:

* Pregnant or lactating women or women with child bearing potential
* Patients with other malignancies except except adequately treated basal cell carcinoma of the skin or in-situ cervix carcinoma
* Active infection or other serious underlying medical condition which would impair the ability of the patient to receive protocol treatment
* Clinical and/or radiological evidence of distant metastases.
* Evidence of pathological fracture
* Prior treatment with an aromatase inhibitor
* Prior administration of any intravenous bisphosphonate during the last year.
* Oral bisphosphonate must be discontinued within 4 weeks of enrollment
* Administration of long-term systemic corticosteroids within the last 12 months (short term steroid treatment is allowed.)
* Prior use of parathyroid hormone treatment for more than 1 week
* Use of any drug known to affect the skeleton (calcitonin, mithramycin, gallium nitrate) within two weeks prior to enrollment
* Abnormal renal function: creatinine clearance must be above 30 ml/min (calculated by Cockroft formula)
* Evidence of metabolic bone disease( Paget's, osteogenesis imperfecta, hyperparathyroidism within the 12 months prior to enrollment)
* Baseline lumbar spine and or total hip Bone Mineral Density T score below -2
* Known hypersensitivity to zoledronic acid
* Psychological, familial, sociologic, or geographic conditions which do not permit medical follow-up and compliance with the study protocol
* White blood cell ≤ 3.0 x 10exp9 /L or granulocytes ≤ 1.5 x 10exp9/L or platelets ≤100 x 10exp9
* Total bilirubin> 1.5 x upper normal limit, SGOT and SGPT > 2.5 x upper normal limit
* Unable to undergo DXA bone density scanning (spine deformity, severe scoliosis, lumbar sacral spine surgery)

Ages: 18 Years to 82 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-09; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
bone mineral density
bone events
renal function
liver function

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Safra, M.D., Study Chair — Tel-Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Soroka University Medical Center, Beersheba
  - Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Safra T, Bernstein-Molho R, Greenberg J, Pelles-Avraham S, Stephansky I, Sarid D, Inbar MJ, Stemmer SM, Geffen DB. The protective effect of zoledronic acid on bone loss in postmenopausal women with early breast cancer treated with sequential tamoxifen and letrozole: a prospective, randomized, phase II trial. Oncology. 2011;81(5-6):298-305. doi: 10.1159/000334456. Epub 2011 Dec 8. PMID 22156381